CLINICAL TRIAL: NCT00578175
Title: Immunogenicity of GlaxoSmithKline Biologicals' MMRV Vaccine (208136) vs. ProQuad®, When Coadministered With Hepatitis A and Pneumococcal Conjugate Vaccines to Children 12-14 Months of Age.
Brief Title: Immunogenicity and Safety of GlaxoSmithKline Biologicals' MMRV Vaccine vs. ProQuad® in Children 12-14 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110058
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Results first posted 2010-08-26 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2016-10

CONDITIONS: Varicella; Rubella; Mumps; Measles
Keywords: Vaccines; Rubella; Varicella Vaccine; Children; Humans; Mumps; Immunogenicity; Safety; Measles; Combined Vaccine
MeSH Terms: conditions — Chickenpox; Rubella; Mumps; Measles | interventions — measles, mumps, rubella, varicella vaccine; Hepatitis A Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Group A (Experimental): Subjects received refrigerator-stored Priorix-Tetra™ (MMRV vaccine 208136 formulation A) co-administered with Havrix® and Prevnar® at Day 0 and a second dose of Havrix® at Day 180
  Interventions: Biological: Priorix-Tetra™ (MMRV vaccine 208136); Biological: Havrix®; Biological: Prevnar®
- Group B (Experimental): Subjects received freezer-stored Priorix-Tetra™ (MMRV vaccine 208136 formulation B) co-administered with Havrix® and Prevnar® at Day 0 and a second dose of Havrix® at Day 180
  Interventions: Biological: Priorix-Tetra™ (MMRV vaccine 208136); Biological: Havrix®; Biological: Prevnar®
- Group C (Active Comparator): Subjects received ProQuad® co-administered with Havrix® and Prevnar® at Day 0 and a second dose of Havrix® at Day 180
  Interventions: Biological: ProQuad®; Biological: Havrix®; Biological: Prevnar®

INTERVENTIONS:
Biological: Priorix-Tetra™ (MMRV vaccine 208136) — One subcutaneous injection.
  Arms: Group A; Group B
Biological: ProQuad® — One subcutaneous injection.
  Arms: Group C
Biological: Havrix® — Two intramuscular injections.
Biological: Prevnar® — One intramuscular injection.

SUMMARY:
The purpose of this observer blinded study is to provide information on vaccine immunogenicity and reactogenicity in comparison with the US standard of care (ProQuad®) when administered with Hepatitis A vaccine and Pneumococcal vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes their parents/guardians can and will comply with the requirements of the protocol.
* Male or female between 12 and 14 months of age at the time of first vaccination.
* Written informed consent obtained from the parent/guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Have previously received 3 doses of 7-valent pneumococcal conjugate vaccine within the first year of life.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol from 30 days prior to vaccination until 42 days after vaccination, except for influenza vaccine.
* Previous vaccination against measles, mumps, rubella and/or varicella.
* Previous vaccination against hepatitis A or receipt of a fourth dose of pneumococcal conjugate vaccine.
* History of measles, mumps, rubella and/or varicella/zoster diseases.
* Known exposure to measles, mumps, rubella and/or varicella/zoster within 30 days prior to the start of the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination, including human immunodeficiency virus infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures. Uncomplicated febrile convulsions are not an exclusion criterion.
* Residence in the same household as the following persons:

  * New-born infants (0-4 weeks of age).
  * Pregnant mother/women with a negative history of chickenpox disease and without recorded vaccination against chickenpox.
  * Pregnant women at or beyond 28 weeks gestation regardless of varicella vaccination status or varicella disease history.
  * Persons with known immunodeficiency.
* Acute disease at the time of enrolment. All vaccines can be administered to persons with a minor illness.
* Administration of polyclonal immunoglobulins and/or any blood products during the six months before entering the study or planned administration during the study period.
* Contra-indications to commercially available vaccines used in this study (Havrix®, Prevnar®, ProQuad®).

Ages: 12 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1851 (Actual)
Dates: Start 2007-11-20; Primary Completion 2009-02-24 (Actual); Study Completion 2009-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (128):
- United States (128):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Buena Park, California
  - GSK Investigational Site, Downey, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Lakewood, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Pleasanton, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Vacaville, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Thornton, Colorado
  - GSK Investigational Site, Westminster, Colorado
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Opa-locka, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Carrollton, Georgia
  - GSK Investigational Site, Dalton, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Tifton, Georgia
  - GSK Investigational Site, Tucker, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Fishers, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, Dubuque, Iowa
  - GSK Investigational Site, Waukee, Iowa
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Topeka, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Springfield, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Portage, Michigan
  - GSK Investigational Site, Richland, Michigan
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Brainerd, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Bridgeton, Missouri
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Whitehouse Station, New Jersey
  - GSK Investigational Site, Johnson City, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Boone, North Carolina
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Sylva, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Minot, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Fairfield, Ohio
  - GSK Investigational Site, Huber Heights, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, East Norriton, Pennsylvania
  - GSK Investigational Site, Kittanning, Pennsylvania
  - GSK Investigational Site, Latrobe, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Sellersville, Pennsylvania
  - GSK Investigational Site, Uniontown, Pennsylvania
  - GSK Investigational Site, Wexford, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Brentwood, Tennessee
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Vienna, Virginia
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, La Crosse, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Blatter MM, Klein NP, Shepard JS, Leonardi M, Shapiro S, Schear M, Mufson MA, Martin JM, Varman M, Grogg S, London A, Cambron P, Douha M, Nicholson O, da Costa C, Innis BL. Immunogenicity and safety of two tetravalent (measles, mumps, rubella, varicella) vaccines coadministered with hepatitis a and pneumococcal conjugate vaccines to children twelve to fourteen months of age. Pediatr Infect Dis J. 2012 Aug;31(8):e133-40. doi: 10.1097/INF.0b013e318259fc8a. PMID 22622699
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110058 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While the total numbers of subjects enrolled in the study was of 1851, the total number of subjects that entered the study was 1783. The remaining 67 subjects received a subject number but no vaccine dose and were therefore excluded from the analysis and group assignment.
Groups:
- Refrigerator-stored Priorix-Tetra Group: Subjects received at Day 0 a single dose of refrigerator-stored Priorix-Tetra subcutaneously in the right upper arm co-administered with a single dose of Havrix and Prevnar intramuscularly in the left and right thigh respectively. At Day 180 they received a second dose of Havrix intramuscularly in the left thigh.
- Freezer-stored Priorix-Tetra Group: Subjects received at Day 0 a single dose of freezer-stored Priorix-Tetra subcutaneously in the right upper arm co-administered with a single dose of Havrix and Prevnar intramuscularly in the left and right thigh respectively. At Day 180 they received a second dose of Havrix intramuscularly in the left thigh.
- Proquad Group: Subjects received at Day 0 a single dose of ProQuad subcutaneously in the right upper arm co-administered with a single dose of Havrix and Prevnar intramuscularly in the left and right thigh respectively. At Day 180 they received a second dose of Havrix intramuscularly.
Period: Overall Study
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Started | 705 | 689 | 389
Completed | 635 | 646 | 365
Not Completed | 70 | 43 | 24
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Other reasons | 70 | 42 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group | Total
Number analyzed (Participants) | 705 | 689 | 389 | 1783
Age, Continuous [Mean (Standard Deviation); unit: months] | 12.3 (0.58) | 12.3 (0.59) | 12.3 (0.61) | 12.3 (0.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 356 | 346 | 186 | 888
  Male | 349 | 343 | 203 | 895

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Seroresponse for Antibodies to Varicella Virus (VZV)
Description: Seroresponse for antibodies to VZV is defined as the appearance post-vaccination of anti-VZV antibodies [concentration greater than or equal to the threshold of 75 milli-international units per milliliter (mIU/mL)] in the serum of subjects below the assay cut-off value of 25 mIU/mL before vaccination.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 622 | 630 | 347
subjects | 355 | 440 | 301

2. Primary Outcome: Concentration of Antibodies to Varicella Virus (VZV)
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 629 | 636 | 352
milli-international units per milliliter | 83.6 [77.0 to 90.8] | 109.9 [102.1 to 118.3] | 164.3 [152.3 to 177.3]

3. Primary Outcome: Number of Subjects With Seroresponse for Antibodies to Mumps Virus
Description: Seroresponse for antibodies to mumps virus is defined as the appearance post-vaccination of anti-mumps virus antibodies [titer greater than or equal to the threshold of 51 Effective Doses (ED50)] in the serum of subjects below the assay cut-off value of 24 ED50 before vaccination.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 532 | 531 | 276
subjects | 491 | 498 | 256

4. Primary Outcome: Number of Subjects With Seroresponse for Antibodies to Measles Virus
Description: Seroresponse for antibodies to measles virus is defined as the appearance post-vaccination of anti-measles virus antibodies [concentration greater than or equal to the threshold of 200 milli-international units per milliliter (mIU/mL)] in the serum of subjects below the assay cut-off value of 150 mIU/mL before vaccination.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Groups:
- Refrigerator-stored Priorix-Tetra Group: Subjects received at Day 0 a single dose of refrigerator-stored Priorix-Tetra subcutaneously in the right upper arm co-administered with a single dose of Havrix and Prevnar intramuscularly in the left and right thigh respectively. At Day 180 they received a second dose of Havrix intramuscularly in the left thigh. .
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 626 | 636 | 350
subjects | 616 | 633 | 342

5. Primary Outcome: Number of Subjects With Seroresponse for Antibodies to Rubella Virus
Description: Seroresponse for antibodies to rubella virus is defined as the appearance post-vaccination of anti-rubella virus antibodies [concentration greater than or equal to the threshold of 10 international units per milliliter (IU/mL)] in the serum of subjects below the assay cut-off value of 4 IU/mL before vaccination.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 628 | 636 | 351
subjects | 616 | 622 | 349

6. Primary Outcome: Concentration of Antibodies to Hepatitis A Virus (HAV)
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 404 | 409 | 227
milli-international units per milliliter | 40.5 [37.1 to 44.2] | 40.3 [37.0 to 44.0] | 40.0 [35.7 to 44.9]

7. Primary Outcome: Concentration of Antibodies to S. Pneumoniae Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
Number analyzed (Participants) | 461 | 468 | 266
micrograms per milliliter (µg/mL)
  S.Pneu.4 (n= 461, 463, 266) | 3.35 [3.10 to 3.63] | 3.31 [3.04 to 3.59] | 3.02 [2.72 to 3.34]
  S.Pneu.6B (n= 460, 464, 265) | 5.65 [5.16 to 6.19] | 5.91 [5.40 to 6.45] | 5.43 [4.90 to 6.02]
  S.Pneu.9V (n=461, 468, 266) | 5.81 [5.37 to 6.29] | 5.66 [5.23 to 6.13] | 5.54 [5.02 to 6.12]
  S.Pneu.14 (n= 460, 465, 266) | 9.71 [8.99 to 10.50] | 9.54 [8.81 to 10.34] | 8.96 [8.07 to 9.95]
  S.Pneu.18C (n= 458, 465, 263) | 5.50 [5.04 to 6.01] | 5.80 [5.30 to 6.34] | 5.51 [4.95 to 6.12]
  S.Pneu.19F (n= 454, 460, 261) | 2.52 [2.32 to 2.74] | 2.52 [2.32 to 2.73] | 2.31 [2.06 to 2.59]
  S.Pneu.23F (n= 459, 464, 266) | 10.10 [9.22 to 11.06] | 10.85 [9.87 to 11.91] | 9.79 [8.65 to 11.07]

8. Secondary Outcome: Antibody Titers to Mumps Virus
Description: Data are expressed as Geometric Mean Titers (GMTs). The titer is the serum dilution giving a 50 percent reduction of the signal compared to a control without serum.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 591 | 601 | 327
titer | 222.4 [202.5 to 244.3] | 224.6 [206.9 to 243.9] | 253.1 [222.7 to 287.7]

9. Secondary Outcome: Concentration of Antibodies to Measles Virus
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-international units per milliliter
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 626 | 636 | 350
milli-international units per milliliter | 4723.1 [4436.4 to 5028.4] | 4650.3 [4430.9 to 4880.5] | 4207.1 [3823.3 to 4629.3]

10. Secondary Outcome: Concentration of Antibodies to Rubella Virus
Description: Concentrations are given as Geometric Mean Concentrations (GMCs).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: International units per milliliter
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 629 | 636 | 352
International units per milliliter | 59.9 [55.9 to 64.1] | 57.9 [54.4 to 61.7] | 71.4 [65.5 to 77.8]

11. Secondary Outcome: Number of Subjects With Vaccine Response to Havrix
Description: Vaccine response to Havrix is defined as the appearance post-vaccination of anti-hepatitis A virus (anti-HAV) antibodies [concentration greater than or equal to 15 milli-international units per milliliter (mIU/mL)] in the serum of subjects seronegative before vaccination (concentration below the assay cut-off value of 15 mIU/mL) or having a 2-fold increase above the pre-vaccination concentration in subjects who were seropositive before vaccination.
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 404 | 409 | 227
subjects | 344 | 345 | 195

12. Secondary Outcome: Number of Subjects With Concentration of Antibodies to S. Pneumoniae Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F Equal or Above the Cut-off Value
Description: Cut-off value assessed include 0.05 micrograms per milliliter (µg/mL).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 461 | 468 | 266
subjects
  Anti-S.Pneu-4 (n= 461, 463, 266) | 461 | 463 | 266
  Anti-S.Pneu-6B (n= 460, 464, 265) | 459 | 463 | 265
  Anti-S.Pneu-9V (n= 461, 468, 266) | 461 | 468 | 266
  Anti-S.Pneu-14 (n= 460, 465, 266) | 460 | 465 | 266
  Anti-S.Pneu-18C (n= 458, 465, 263) | 458 | 465 | 263
  Anti-S.Pneu-19F (n= 454, 460, 261) | 454 | 460 | 261
  Anti-S.Pneu-23F (n= 459, 464, 266) | 459 | 464 | 266

13. Secondary Outcome: Number of Subjects With Concentration of Antibodies to S. Pneumoniae Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F Equal or Above the Cut-off Value
Description: Cut-off value assessed include 0.2 micrograms per milliliter (µg/mL).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 461 | 468 | 266
subjects
  Anti-S.Pneu-4 (n= 461, 463, 266) | 461 | 463 | 266
  Anti-S.Pneu-6B (n= 460, 464, 265) | 458 | 460 | 265
  Anti-S.Pneu-9V (n= 461, 468, 266) | 461 | 468 | 266
  Anti-S.Pneu-14 (n= 460, 465, 266) | 460 | 465 | 266
  Anti-S.Pneu-18C (n= 458, 465, 263) | 458 | 464 | 263
  Anti-S.Pneu-19F (n= 454, 460, 261) | 451 | 459 | 259
  Anti-S.Pneu-23F (n= 459, 464, 266) | 459 | 464 | 266

14. Secondary Outcome: Number of Subjects With Concentration of Antibodies to S. Pneumoniae Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F Equal or Above the Cut-off Value
Description: Cut-off value assessed include 0.5 micrograms per milliliter (µg/mL).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 461 | 468 | 266
subjects
  Anti-S.Pneu-4 (n= 461, 463, 266) | 456 | 459 | 265
  Anti-S.Pneu-6B (n= 460, 464, 265) | 453 | 459 | 264
  Anti-S.Pneu-9V (n= 461, 468, 266) | 459 | 466 | 266
  Anti-S.Pneu-14 (n= 460, 465, 266) | 459 | 464 | 266
  Anti-S.Pneu-18C (n= 458, 465, 263) | 458 | 463 | 263
  Anti-S.Pneu-19F (n= 454, 460, 261) | 431 | 448 | 249
  Anti-S.Pneu-23F (n= 459, 464, 266) | 458 | 462 | 266

15. Secondary Outcome: Number of Subjects With Concentration of Antibodies to S. Pneumoniae Serotypes 4, 6B, 9V, 14, 18C, 19F and 23F Equal or Above the Cut-off Value
Description: Cut-off value assessed include 1.0 micrograms per milliliter (µg/mL).
Time Frame: At Day 42 after vaccination
Population: Analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 461 | 468 | 266
subjects
  Anti-S.Pneu-4 (n= 461, 463, 266) | 437 | 423 | 249
  Anti-S.Pneu-6B (n= 460, 464, 265) | 442 | 453 | 259
  Anti-S.Pneu-9V (n= 461, 468, 266) | 450 | 459 | 265
  Anti-S.Pneu-14 (n= 460, 465, 266) | 458 | 463 | 266
  Anti-S.Pneu-18C (n= 458, 465, 263) | 446 | 455 | 259
  Anti-S.Pneu-19F (n= 454, 460, 261) | 390 | 390 | 214
  Anti-S.Pneu-23F (n= 459, 464, 266) | 446 | 458 | 265

16. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling.
Time Frame: During the 4 day follow up period following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 673 | 666 | 378
subjects
  Pain | 136 | 114 | 65
  Redness | 111 | 120 | 54
  Swelling | 50 | 49 | 21

17. Secondary Outcome: Number of Subjects Reporting Fever ≥ 38.0°C/100.4°F and > 39.5°C/103.1°F During the 15-day Follow up Period After Vaccination
Description: Fever was measured rectally.
Time Frame: During the 15-day follow-up period following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 676 | 668 | 379
subjects
  ≥ 38.0°C/100.4°F | 248 | 241 | 120
  > 39.5°C/103.1°F | 33 | 48 | 14

18. Secondary Outcome: Number of Subjects Reporting Fever ≥ 38.0°C/100.4°F and > 39.5°C/103.1°F During the 43-day Follow-up Period After Vaccination
Description: Fever was measured rectally.
Time Frame: During the 43-day follow-up period following vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 676 | 668 | 379
subjects
  ≥ 38.0°C/100.4°F | 312 | 301 | 162
  > 39.5°C/103.1°F | 52 | 71 | 24

19. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Measles/Rubella-like Rash
Time Frame: During the 43-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 676 | 668 | 379
subjects | 37 | 25 | 15

20. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Varicella-like Rash
Time Frame: During the 43-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 676 | 668 | 379
subjects | 10 | 9 | 6

21. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Parotid/Salivary Gland Swelling
Time Frame: During the 43-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 676 | 668 | 379
subjects | 14 | 7 | 5

22. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events and Medically-attended Adverse Events (Excluding Rash and Parotid/Salivary Gland Swelling)
Description: Unsolicited adverse event covers any adverse event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Medically-attended adverse event covers any adverse event which received medical attention. Medical attention is defined as hospitalization, an emergency room visit or a visit to or from medical personnel.
Time Frame: During the 43-day follow-up period after vaccination
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 705 | 689 | 389
subjects
  Unsolicited adverse events | 338 | 332 | 191
  Medically-attended adverse events | 217 | 213 | 124

23. Secondary Outcome: Number of Subjects Reporting New Onset Chronic Illnesses and Conditions Prompting Emergency Room Visits
Description: New onset chronic illnesses include autoimmune disorders, asthma, type I diabetes and allergies.
Time Frame: For approximately 6 months (Day 0-180)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 705 | 689 | 389
subjects
  New onsets of chronic diseases | 11 | 11 | 7
  Emergency room visits | 63 | 63 | 44

24. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: For approximately 6 months (Day 0-180)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | ProQuad Group
Number analyzed (Participants) | 705 | 689 | 389
subjects | 14 | 20 | 7

ADVERSE EVENTS:
Time Frame: Solicited local AEs: during 4-day follow-up period after vaccination. Solicited general & Unsolicited AEs: during 43-day follow-up period after vaccination. SAEs: during the entire study period (approximately 6 months; Day 0 to Day 180).
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available.
  Events collected by non-systematic method are reported for the Total Vaccinated Cohort.
Arm/Group | Refrigerator-stored Priorix-Tetra Group | Freezer-stored Priorix-Tetra Group | Proquad Group
All-Cause Mortality (participants affected / at risk) | 0/705 | 0/689 | 0/389
Serious Adverse Events (participants affected / at risk) | 14/705 | 20/689 | 7/389
Other Adverse Events (participants affected / at risk) | 547/705 | 541/689 | 297/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Refrigerator-stored Priorix-Tetra Group (N=705) | Freezer-stored Priorix-Tetra Group (N=689) | Proquad Group (N=389)
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 2 | 0
Groin abscess (Infections and infestations) | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0
Abscess (Infections and infestations) | 0 | 1 | 0
Accidental drug intake by child (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Autism spectrum disorder (Psychiatric disorders) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Croup infectious (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Hpoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Primitive neuroectodermal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Refrigerator-stored Priorix-Tetra Group (N=705) | Freezer-stored Priorix-Tetra Group (N=689) | Proquad Group (N=389)
Pain (General disorders) | 136/673 | 114/666 | 65/378
Redness (General disorders) | 111/673 | 120/666 | 54/378
Swelling (General disorders) | 50/673 | 49/666 | 21/378
Fever (General disorders) | 312/676 | 302/668 | 163/379
Rash (General disorders) | 221/676 | 219/668 | 128/379
Otitis media (Infections and infestations) | 71 | 62 | 34
Uper respiratory tract infection (Infections and infestations) | 49 | 58 | 42
Teething (Gastrointestinal disorders) | 42 | 53 | 28
Diarrhoea (Gastrointestinal disorders) | 37 | 46 | 29
Irritability (General disorders) | 25 | 35 | 20
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 29 | 21 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.